CLINICAL TRIAL: NCT01859156
Title: End-Tidal Carbon Dioxide as a Measure of Carboxyhemoglobin in Carbon Monoxide
Brief Title: End-Tidal Carbon Dioxide as a Measure of Carboxyhemoglobin in Carbon Monoxide Poisoning
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 06-2713
Record Dates: First submitted 2013-05-08; First posted 2013-05-21 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Carbon Monoxide Exposure
Keywords: Carbon Monoxide; Carboxyhemoglobin; End-tidal carbon dioxide; Capnography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Carbon Monoxide Exposure

SUMMARY:
The purpose of this study is to determine whether a relationship exists between EtCO2 and carboxyhemoglobin levels in carbon monoxide exposure. Our hypothesis is that a liner relationship exists between EtCO2 and carboxyhemoglobin in carbon monoxide poisoning.

ELIGIBILITY:
Inclusion Criteria:

* Carbon monoxide exposure

Exclusion Criteria:

* Less than 18 years old
* Suicide attempt
* Unable to provide informed consent
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department at an urban county hospital.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2006-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
EtCO2 | Immediately upon study enrollment, an average time of 30 minutes post arrival to the hospital.
  The EtCO2 level is measured by capnography and compared to the carboxyhemoglobin level.

CONTACTS AND LOCATIONS:
Overall Officials: James R Miner, MD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States